CLINICAL TRIAL: NCT00368693
Title: Pivotal Study to Evaluate the Efficacy and Safety of Dermal - Living Skin Replacement (Dermal - LSR) in the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Efficacy and Safety Study of Dermal-Living Skin Replacement to Treat Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to low enrollment.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Apopharma RS03-2004; VA File #05-08-00364
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dermal - Living Skin Replacement (Dermal-LSR) — The only experimental procedure is the application of the study device, Dermal - Living Skin Replacement (Dermal - LSR), to the foot ulcer. All others are regular or standard procedures. Dermal - LSR is a gel containing living human skin cells. This gel is applied directly to ulcers to help repair the skin. The cells used in this study device have come from one foreskin (skin covering the tip of the penis) taken from a baby boy shortly after his birth for reasons unrelated to this study. All cells that will be used have been tested to be healthy and safe. The amount of the study device you will receive depends on the size of your ulcer at each treatment visit. You will receive less than a 1/4 teaspoon of Dermal - LSR for about every dime-size area of your ulcer as measured and calculated by the research investigator.

SUMMARY:
The purpose of this study is to test the efficacy and side effects, if any, of Dermal - LSR combined with standard treatment. We hypothesize the treatment will provide beneficial results for diabetic patients suffering foot ulcers.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, open-label, multi-center study will test the efficacy of Dermal - Living Skin Replacement (Dermal - LSR) plus standard of care treatment against solely the standard of care treatment on participants with diabetic foot ulcers.

The purpose of this study is to test Dermal - LSR combined with standard treatment. We want to see how well it works and the number and types of side effects, if any. We hope to learn more about how to heal diabetic foot ulcers better.

You will:

* be interviewed and examined
* have weekly clinic visits
* have blood drawn
* have the ulcer photographed
* wear a walking boot to reduce pressure on the ulcer

ELIGIBILITY:
Inclusion Criteria:

* Have Type I or Type II diabetes
* Signed informed consent obtained from subject or legal guardian/representative prior to the first study intervention.
* Age ≥ 18 and < 85 years old at the time the informed consent is signed.
* Subjects will have a diabetic ulcer on the lower extremity, with the ulcer having all of the following characteristics:

  1. Full-thickness plantar ulcers (fore and mid foot only);
  2. Non-infected as determined by clinical assessment;
  3. Neuropathic as determined by monofilament assessment;
  4. Area ≥ 1.0 cm2 ≤ 25.0 cm2 post-debridement;
  5. Has been present for at least 8 weeks under a physician's observation at the time of enrollment;
  6. Extends through the dermis but without tendon, muscle, capsule or bone exposure.
* Subjects will have only one diabetic foot ulcer on the target limb.
* Subjects will have either insulin-dependent or non-insulin-dependent diabetes mellitus (Type I or Type II, respectively) with a HbA1C value in the range of 6% to 12%.
* The ulcer bed at the time of enrollment must be free of all necrotic and infected soft and bony tissue as determined by clinical examination (no evidence of probing to bone) and by X-ray films.
* Ankle-brachial systolic pressure index between 0.7 and 1.3. If the value is > 1.3, then a transcutaneous partial pressure of oxygen (TcPO2) of ≥ 40 mmHg OR a toe pressure of ≥ 50 mmHg must be obtained for subject to be eligible.
* Female subjects must have a negative serum pregnancy test prior to the first treatment.

Exclusion Criteria:

* Known or suspected disease of the immune system currently under investigation, other than Diabetes Mellitus.
* Active or untreated malignancy or active, uncontrolled connective tissue disease.
* Treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or corticosteroids less than 30 days before enrollment.
* Presence of necrosis, purulence or sinus tracts that cannot be removed by treatment.
* Has undergone a revascularization procedure aimed at increasing blood flow in the treatment target limb < 4 weeks prior to enrollment.
* Active febrile illness (fever ≥ 38.0 ºC p.o.).
* Renal or liver impairment as indicated by serum creatinine levels and liver function tests three or more times higher than the normal values.
* Osteomyelitis diagnosed by exposed bone and by radiological investigations.
* Subject has an active Charcot as determined by the clinical examination (new local pain, evidence of swelling and warmth).
* Subjects who refuse or who are unable to participate in all screening procedures, or to comply with the requirements of the study.
* Use of other investigational products at the time of enrollment or during the study.
* The use of any topical treatments, other than SOC, in or on the surface of the target ulcer at the time of enrollment.
* Subjects who have been enrolled in any investigational clinical trial within 30 days of the screening visit.
* Currently pregnant or lactating, or planning a pregnancy to occur during the study period.
* Known allergic reactions, including dermatological hypersensitivity, to any study product components.
* Recent or current history of alcohol or drug abuse.
* Subjects who, in the opinion of the Investigator, represent poor medical, psychological or psychiatric risks for whom therapy with an investigational product would be unwise.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Complete ulcer closure will be defined as complete re-epithelialization without the presence of any callus and/or exudate. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roslyn R Isseroff, M.D., Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - VA Medical Center, Mather, California
  - University of California, Davis Medical Center Department of Dermatology, Sacramento, California

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical